CLINICAL TRIAL: NCT00234091
Title: An Open Label, Randomized Study to Compare Antiretroviral Therapy (ART) Initiation When CD4 is Between 15% to 24% to ART Initiation When CD4 Falls Below 15% in Children With HIV Infection and Moderate Immune Suppression
Brief Title: When to Start Anti-HIV Drugs in Children Infected With HIV (The PREDICT Study)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Comprehensive International Program of Research on AIDS (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CIPRA TH001; PREDICT; 10409 (Registry Identifier: DAIDS ES)
Record Dates: First submitted 2005-10-04; First posted 2005-10-06 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-12

CONDITIONS: HIV Infections
Keywords: Treatment Naive; Treatment Initiation; Infant; Preschool Child; Child; Zidovudine; AZT; Retrovir; 3TC; Lamivudine; Epivir; Nevirapine; NVP; Viramune; Efavirenz; EFV; Sustiva; Lopinavir/Ritonavir; LPV/r; Kaletra; Nelfinavir; NFV; Viracept; ABC; Abacavir; Ziagen
MeSH Terms: conditions — HIV Infections | interventions — abacavir; efavirenz; Lamivudine; Lopinavir; Nelfinavir; Nevirapine; Zidovudine

ARMS (2):
- 1 (Active Comparator): Immediate treatment; individuals receive HAART on Day 1 of the study
  Interventions: Drug: Abacavir; Drug: Efavirenz; Drug: Lamivudine; Drug: Lopinavir/Ritonavir; Drug: Nelfinavir; Drug: Nevirapine; Drug: Zidovudine
- 2 (Active Comparator): Delayed treatment; individuals receive HAART if their CD4 percentage falls below 15 percentage OR if they develop a CDC category C illness
  Interventions: Drug: Abacavir; Drug: Efavirenz; Drug: Lamivudine; Drug: Lopinavir/Ritonavir; Drug: Nelfinavir; Drug: Nevirapine; Drug: Zidovudine

INTERVENTIONS:
Drug: Abacavir — 8 mg/kg (up to 300 mg/dose) take orally twice daily
Drug: Efavirenz — 200 to 600 mg taken orally once daily
Drug: Lamivudine — 4 mg/kg (up to 150 mg/dose) taken orally twice daily
Drug: Lopinavir/Ritonavir — 230 mg/57.5 mg/m^2 body surface area taken orally twice daily with food
Drug: Nelfinavir — 45-55 mg/kg taken orally twice daily with food
Drug: Nevirapine — 120 mg/m^2 once daily for first 14 days, tehn 200 mg/m^2 (up to 400 mg/day) twice daily
Drug: Zidovudine — 180-240 mg/m^2 every 12 hours (up to 300 mg/dose)

SUMMARY:
The purpose of this study is to determine when HIV infected children should begin taking anti-HIV medications in order to improve both patient quality of life and survival.

DETAILED DESCRIPTION:
The use of highly active antiretroviral therapy (HAART) has resulted in a significant reduction in AIDS-related deaths and complications among adults and adolescents. However, the medical management of HIV infected children remains challenging. Access to HIV treatment is limited and early treatment initiation can cause serious complications. Since there is currently no cure for HIV, a balance between treating the disease and maintaining quality of life must be weighed carefully. An evaluation to determine the appropriate time to initiate HAART is necessary to improve both quality of life and survival for HIV infected children.

This study will last 144 weeks. All participants will have a CD4 percentage (CD4%) between 15% and 24% and will be randomly assigned to either receive immediate or delayed HAART. The HAART regimen will consist of two nucleoside reverse transcriptase inhibitors, zidovudine and lamivudine. In addition, participants will also receive either one non-nucleoside reverse transcriptase inhibitor, nevirapine or efavirenz, or one protease inhibitor, ritonavir-boosted lopinavir or nelfinavir. Abacavir will replace zidovudine or lamivudine if participants experience toxicity to the regimen. Participants in the immediate treatment arm will receive HAART on Day 1 of the study regardless of their CD4%. Participants in the delayed treatment arm will receive HAART if their CD4% falls below 15 or if they develop a CDC Category C illness.

Study visits will occur every 4 weeks for the first 12 weeks and then every 12 weeks until the end of the study. Blood collection, physical exams, and medical and medication history reviews will occur at all visits. Adherence, quality of life, and lipodystrophy assessments will occur every 12 weeks for participants on HAART. Participants will be encouraged to enroll in a related substudy to examine the neurodevelopment of HIV infected children.

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infected
* Antiretroviral naive, defined as never receiving anti-HIV medications, receiving them for less than 7 days, or only receiving them to prevent mother-to-child transmission (MTCT)
* CD4% between 15 and 24 within 30 days prior to study entry
* CDC pediatric clinical classification A or B
* Parent or guardian willing to provide informed consent and willing to follow all study procedures and requirements

Exclusion Criteria:

* Use of systemic chemotherapy, immunomodulators, HIV vaccines, immune globulin, interleukins, or interferons within 30 days prior to study entry
* Active AIDS-defining illnesses (CDC Category C) within 30 days prior to study entry
* Certain abnormal laboratory values
* Known kidney disease
* Known allergy or sensitivity to study drugs
* Require certain medications
* Pregnancy

Ages: 1 Year to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2006-04; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
AIDS-free survival | Week 144

SECONDARY OUTCOMES:
Direct and indirect cost of treatment per patient | Week 144
Number and duration of hospitalizations | throughout study
Time to and number of Grades 3 or 4 HAART-related toxicity and intolerance | throughout study
Number of HAART regimen changes | throughout study
Number of Grades 1 or 2 infectious episodes | throughout study
Number of courses of antibiotics used | throughout study
Number of HIV-related clinical events | throughout study
Virologic failure, defined as HIV viral load of 1000 copies/ml | Week 24 after HAART initiation
Presence of a resistance mutation in participants with virologic failure | throughout study
Change of growth in Z scores | study entry to Week 144
Change in CD4% and time-weighted average change | study entry and Week 144
CD4 less than 10% | Week 144
Average scores of the child's quality of life over time | Week 144
Percentage adherence to HAART over time by pill count/weighing liquid medication bottles, self report, and questionnaire | throughout study
Presence of iron deficiency anemia | study entry and Weeks 24, 48, 72, 96, 120, and 144
HIV viral sequence | study entry and treatment failure
HIV viral replication capacity | throughout study
Cytotoxic T-cell (CTL) response | throughout study
Percentage of different T-cell subsets | study entry and Weeks 48, 96, and 144

CONTACTS AND LOCATIONS:
Overall Officials: Kiat Ruxrungtham, MD, MPH, Study Chair — Department of Medicine at Chulalongkorn University, Bangkok, Thailand; Saphonn Vonthanak, MD, PhD, Study Chair — National Center for HIV/AIDS Dermatology and STDs, Phnom Penh, Cambodia
Locations (9):
- Cambodia (2):
  - National Pediatric Hosp., Cambodia CIPRA CRS, Phnom Penh
  - Social Health Clinic, Cambodia CIPRA CRS, Phnom Penh
- Thailand (7):
  - Hiv-Nat Cipra Crs, Pathumwan, Bangkok
  - Chiang Rai Regional Hosp. CIPRA CRS, Muang, Changwat Chiang Rai
  - Prapokklao Hosp. CIPRA CRS, Chanthaburi
  - Nakornping Hosp. CIPRA CRS, Chiang Mai
  - Queen Savang Vadhana Memorial Hosp. CIPRA CRS, Chon Buri
  - Srinagarind Hosp. CIPRA CRS, Khon Kaen
  - Bamrasnaradura Institute CIPRA CRS, Nonthaburi

REFERENCES:
- [Background] Lindsey JC, Malee KM, Brouwers P, Hughes MD; PACTG 219C Study Team. Neurodevelopmental functioning in HIV-infected infants and young children before and after the introduction of protease inhibitor-based highly active antiretroviral therapy. Pediatrics. 2007 Mar;119(3):e681-93. doi: 10.1542/peds.2006-1145. Epub 2007 Feb 12. PMID 17296781
- [Background] Nikolic-Djokic D, Essajee S, Rigaud M, Kaul A, Chandwani S, Hoover W, Lawrence R, Pollack H, Sitnitskaya Y, Hagmann S, Jean-Philippe P, Chen SH, Radding J, Krasinski K, Borkowsky W. Immunoreconstitution in children receiving highly active antiretroviral therapy depends on the CD4 cell percentage at baseline. J Infect Dis. 2002 Feb 1;185(3):290-8. doi: 10.1086/338567. Epub 2002 Jan 8. PMID 11807710
- [Background] Puthanakit T, Aurpibul L, Oberdorfer P, Akarathum N, Kanjananit S, Wannarit P, Sirisanthana T, Sirisanthana V. Hospitalization and mortality among HIV-infected children after receiving highly active antiretroviral therapy. Clin Infect Dis. 2007 Feb 15;44(4):599-604. doi: 10.1086/510489. Epub 2007 Jan 9. PMID 17243067
- [Background] Walker AS, Doerholt K, Sharland M, Gibb DM; Collaborative HIV Paediatric Study (CHIPS) Steering Committee. Response to highly active antiretroviral therapy varies with age: the UK and Ireland Collaborative HIV Paediatric Study. AIDS. 2004 Sep 24;18(14):1915-24. doi: 10.1097/00002030-200409240-00007. PMID 15353977
- [Derived] Paul RH, Cho KS, Belden AC, Mellins CA, Malee KM, Robbins RN, Salminen LE, Kerr SJ, Adhikari B, Garcia-Egan PM, Sophonphan J, Aurpibul L, Thongpibul K, Kosalaraksa P, Kanjanavanit S, Ngampiyaskul C, Wongsawat J, Vonthanak S, Suwanlerk T, Valcour VG, Preston-Campbell RN, Bolzenious JD, Robb ML, Ananworanich J, Puthanakit T; PREDICT Study Group. Machine-learning classification of neurocognitive performance in children with perinatal HIV initiating de novo antiretroviral therapy. AIDS. 2020 Apr 1;34(5):737-748. doi: 10.1097/QAD.0000000000002471. PMID 31895148
- [Derived] Paul R, Apornpong T, Prasitsuebsai W, Puthanakit T, Saphonn V, Aurpibul L, Kosalaraksa P, Kanjanavanit S, Luesomboon W, Ngampiyaskul C, Suwanlerk T, Chettra K, Shearer WT, Valcour V, Ananworanich J, Kerr S. Cognition, Emotional Health, and Immunological Markers in Children With Long-Term Nonprogressive HIV. J Acquir Immune Defic Syndr. 2018 Apr 1;77(4):417-426. doi: 10.1097/QAI.0000000000001619. PMID 29303843
- [Derived] Paul R, Prasitsuebsai W, Jahanshad N, Puthanakit T, Thompson P, Aurpibul L, Hansudewechakul R, Kosalaraksa P, Kanjanavanit S, Ngampiyaskul C, Luesomboon W, Lerdlum S, Pothisri M, Visrutaratna P, Valcour V, Nir TM, Saremi A, Kerr S, Ananworanich J; Pediatric Randomized Early versus Deferred Initiation in Cambodia and Thailand (PREDICT) Study Group. Structural Neuroimaging and Neuropsychologic Signatures in Children With Vertically Acquired HIV. Pediatr Infect Dis J. 2018 Jul;37(7):662-668. doi: 10.1097/INF.0000000000001852. PMID 29200184
- [Derived] Bunupuradah T, Hansudewechakul R, Kosalaraksa P, Ngampiyaskul C, Kanjanavanit S, Wongsawat J, Luesomboon W, Sophonphan J, Puthanakit T, Ruxrungtham K, Shearer WT, Ananworanich J; PREDICT study group. HLA-DRB1454 and predictors of new-onset asthma in HIV-infected Thai children. Clin Immunol. 2015 Mar;157(1):26-9. doi: 10.1016/j.clim.2014.12.006. Epub 2014 Dec 26. No abstract available. PMID 25546395
- [Derived] Intasan J, Bunupuradah T, Vonthanak S, Kosalaraksa P, Hansudewechakul R, Kanjanavanit S, Ngampiyaskul C, Wongsawat J, Luesomboon W, Apornpong T, Kerr S, Ananworanich J, Puthanakit T; PREDICT Study Group. Comparison of adherence monitoring tools and correlation to virologic failure in a pediatric HIV clinical trial. AIDS Patient Care STDS. 2014 Jun;28(6):296-302. doi: 10.1089/apc.2013.0276. PMID 24901463
- [Derived] Puthanakit T, Saphonn V, Ananworanich J, Kosalaraksa P, Hansudewechakul R, Vibol U, Kerr SJ, Kanjanavanit S, Ngampiyaskul C, Wongsawat J, Luesomboon W, Ngo-Giang-Huong N, Chettra K, Cheunyam T, Suwarnlerk T, Ubolyam S, Shearer WT, Paul R, Mofenson LM, Fox L, Law MG, Cooper DA, Phanuphak P, Vun MC, Ruxrungtham K; PREDICT Study Group. Early versus deferred antiretroviral therapy for children older than 1 year infected with HIV (PREDICT): a multicentre, randomised, open-label trial. Lancet Infect Dis. 2012 Dec;12(12):933-41. doi: 10.1016/S1473-3099(12)70242-6. Epub 2012 Oct 9. PMID 23059199
- [Derived] Kosalaraksa P, Bunupuradah T, Vonthanak S, Wiangnon S, Hansudewechakul R, Vibol U, Kanjanavanit S, Ngampiyaskul C, Wongsawat J, Luesomboon W, Lumbiganon P, Sopa B, Apornpong T, Chuenyam T, Cooper DA, Ruxrungtham K, Ananworanich J, Puthanakit T. Prevalence of anemia and underlying iron status in naive antiretroviral therapy HIV-infected children with moderate immune suppression. AIDS Res Hum Retroviruses. 2012 Dec;28(12):1679-86. doi: 10.1089/AID.2011.0373. Epub 2012 Jul 25. PMID 22734817
- [Derived] Bunupuradah T, Ubolyam S, Hansudewechakul R, Kosalaraksa P, Ngampiyaskul C, Kanjanavanit S, Wongsawat J, Luesomboon W, Pinyakorn S, Kerr S, Ananworanich J, Chomtho S, van der Lugt J, Luplertlop N, Ruxrungtham K, Puthanakit T; PREDICT study group. Correlation of selenium and zinc levels to antiretroviral treatment outcomes in Thai HIV-infected children without severe HIV symptoms. Eur J Clin Nutr. 2012 Aug;66(8):900-5. doi: 10.1038/ejcn.2012.57. Epub 2012 Jun 20. PMID 22713768
- [Derived] Kanjanavanit S, Puthanakit T, Vibol U, Kosalaraksa P, Hansudewechakul R, Ngampiyasakul C, Wongsawat J, Luesomboon W, Wongsabut J, Mahanontharit A, Suwanlerk T, Saphonn V, Ananworanich J, Ruxrungtham K; PREDICT study group. High prevalence of lipid abnormalities among antiretroviral-naive HIV-infected Asian children with mild-to-moderate immunosuppression. Antivir Ther. 2011;16(8):1351-5. doi: 10.3851/IMP1897. PMID 22155918
- [Derived] Bunupuradah T, Puthanakit T, Kosalaraksa P, Kerr SJ, Kariminia A, Hansudewechakul R, Kanjanavanit S, Ngampiyaskul C, Wongsawat J, Luesomboon W, Chuenyam T, Vonthanak S, Vun MC, Vibol U, Vannary B, Ruxrungtham K, Ananworanich J; PREDICT Study Group. Poor quality of life among untreated Thai and Cambodian children without severe HIV symptoms. AIDS Care. 2012;24(1):30-8. doi: 10.1080/09540121.2011.592815. Epub 2011 Jul 21. PMID 21777076
- [Derived] Ananworanich J, Apornpong T, Kosalaraksa P, Jaimulwong T, Hansudewechakul R, Pancharoen C, Bunupuradah T, Chandara M, Puthanakit T, Ngampiyasakul C, Wongsawat J, Kanjanavanit S, Luesomboon W, Klangsinsirikul P, Ngo-Giang-Huong N, Kerr SJ, Ubolyam S, Mengthaisong T, Gelman RS, Pattanapanyasat K, Saphonn V, Ruxrungtham K, Shearer WT; PREDICT Study Group. Characteristics of lymphocyte subsets in HIV-infected, long-term nonprogressor, and healthy Asian children through 12 years of age. J Allergy Clin Immunol. 2010 Dec;126(6):1294-301.e10. doi: 10.1016/j.jaci.2010.09.038. PMID 21134574
- [Derived] Wongsawat J, Puthanakit T, Kanjanavanit S, Hansudewechakul R, Ngampiyaskul C, Kerr SJ, Ubolyam S, Suwanlerk T, Kosalaraksa P, Luesomboon W, Ngo-Giang-Huong N, Chandara M, Saphonn V, Ruxrungtham K, Ananworanich J; PREDICT Study Group. CD4 cell count criteria to determine when to initiate antiretroviral therapy in human immunodeficiency virus-infected children. Pediatr Infect Dis J. 2010 Oct;29(10):966-8. doi: 10.1097/INF.0b013e3181e0554c. PMID 20418798
- See also: Click here for more information about the HIV Netherlands Australia Thailand Research Collaboration (HIV-NAT) — http://www.hivnat.org